## **DEPARTMENT OF PSYCHIATRY**

NEUROSCIENCES BUILDING WARNEFORD HOSPITAL OXFORD OX3 7JX, U.K. www.psych.ox.ac.uk



TEL. (Direct) 01865 618313 Email: susannah.murphy@psych.ox.ac.uk

## INFORMED CONSENT FORM

**Title of Project:** The effect of seven day prucal opride administration on emotional

processing in healthy volunteers

**Researcher:** Dr Susannah Murphy, Principal Investigator

Please initial the box next to each statement

The purpose of this study is to investigate the effects of prucal opride on emotional processing and neural activity, comparing the effects of the drug with placebo.

University of Oxford Central University Research Ethics Committee: R57219/RE001

| I confirm that I have read and understood the information sheet dated (Version) for the above study. I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily. |
|---|
| I understand that my participation is voluntary and that I am free to withdraw at any time, without giving reason, and without any adverse consequences or academic penalty. |
| I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. |
| I have been advised as to what I need to do for this research (especially with regard to drug intake) and I agree to follow the instructions given to me. |
| I understand that research data and scan images collected during the study may<br>be looked at by designated individuals from the University of Oxford where it is<br>relevant to my taking part in this study. I give permission for these individuals to<br>access my data. |
| I understand who will have access to personal data provided, how the data will be stored and what will happen to the data at the end of the project. |

| I consent to answering screening questions, including questions about my physical and mental health, to confirm my eligibility to take part. |
|---|
| I understand that this project has been reviewed, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. |
| I understand how this research will be written up and published. |
| I understand how to raise a concern or make a complaint. |
| I understand that all information will be kept strictly confidential except in the rare circumstance in which it is judged that I, or someone else, is at immediate risk of serious harm. |
| I understand that the MRI scans in this study are for research and they are not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will be informed if a doctor thinks this is medically important such that the finding has clear implications for my current or future health. |
| I agree for research data collected in this study to be given to researchers, including those working outside of the EU, to be used in other research studies. I give permission for data from this study to be used in publication. I understand that any data and/or brain images of me that leave the Department will be fully anonymised so that I cannot be identified. |
| I understand that I have been advised not to drink alcohol or carry out activities requiring full alertness (such as driving) during the week of drug/placebo administration if I am aware of any impairment. |
| I agree to take part in this study. |
| (Optional) I agree to being contacted about future studies for which I might be suitable, without any commitment to take part. I agree to my contact details being retained from my screening form, and entered into a database, for this purpose. |

| Name of participant: | |
|----------------------------------------------|-------|
| Signature: | Date: |
| Name of person taking consent: | |
| Signature: | Date: |
| One copy for participant, one for researcher | |